CLINICAL TRIAL: NCT02945098
Title: Kinesio Taping® Does Not Interfere in Muscle Damage Response Induced by Eccentric Exercise: a Randomized Controlled Trial
Brief Title: Kinesio Taping in Muscle Damage Response Induced by Eccentric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Professor of Physiotherapy, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LAPERN09
Record Dates: First submitted 2016-10-23; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Bandages; Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): No intervention. Remained five minutes at rest.
- Placebo group (Placebo Comparator): Apply Kinesio Taping without tension.
  Interventions: Other: Placebo Kinesio Taping
- KT group (Experimental): Apply Kinesio Taping application with tension.
  Interventions: Other: Kinesio Taping

INTERVENTIONS:
Other: Kinesio Taping — Kinesio Taping application with tension (Kinesio Tex Gold®, Japan) in the anterior region of the non-dominant arm.
  Other Names: Functional elastic tape
  Arms: KT group
Other: Placebo Kinesio Taping — Kinesio Taping application without tension (Kinesio Tex Gold®, Japan) in the anterior region of the non-dominant arm.
  Other Names: Placebo functional elastic tape
  Arms: Placebo group

SUMMARY:
Sixty volunteers with a mean age of 21,8 ± 2,6 years participated in this study, randomly distributed into one of the following groups: control, Kinesio taping group with tension in the anterior arm region and Kinesio taping group without tension in the same region. All subjects underwent an eccentric exercise protocol and three evaluations: before the protocol, immediately after and 48h after protocol. The following variables were analyzed: sensation of pain as the primary outcome; peak torque normalized by body weight; average peak torque; total work and average power, using an isokinetic dynamometer. In addition, muscle activation amplitude (Root Mean Square) and median frequency were recorded using surface electromyography.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 28 years;
* BMI below 30;
* Practicing recreational physical activity at least three times a week without training at a competitive level;
* Exhibiting shoulder joint, elbow and non-dominant hand integrity;
* Do not having a history of osteo-myoarticular injuries in the assessed limb in the last 6 months.

Exclusion Criteria:

* Does not run the tests properly;
* Be allergic to tape test;
* Does not attend all assessments.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | Change from baseline in visual analogue scale at one hour and three days

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No